CLINICAL TRIAL: NCT03501888
Title: A Single Blind Randomized Controlled Trial Comparing Cognitive Behavior Group Therapy and Individual Cognitive Behavioural Therapy for Patients With Psychoses
Brief Title: Cognitive Behavior Therapy for Patients With Psychoses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Helena Fatouros-Bergman, Pricipal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karolinska Inst
Record Dates: First submitted 2017-01-30; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Acceptance and Commitment Therapy; ACT; Cognitive Behavior Therapy; CBT; Schizophrenia; Psychoses
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (CBT) (Active Comparator): CBT: individually, ca 18 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Acceptance and Commitment Therapy (ACT) (Active Comparator): ACT: given in a group setting: ca 18 weeks.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — 18 sessions of individual treatment, no manual.
  Other Names: CBT
  Arms: Cognitive Behavior Therapy (CBT)
Behavioral: Acceptance and Commitment Therapy — 18 sessions of group treatment, manual based.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy (ACT)

SUMMARY:
Patients with psychoses are randomized either to group treatment (ACT) or individual CBT for 18 sessions.

DETAILED DESCRIPTION:
Since patients in the early stage of the illness seem to benefit more from CBT than patients with chronic conditions the present research will focus on patients with psychosis at the early stages of their illness. Patients with first episode psychosis from the Northern Stockholm Psychiatry (Midhagen) and the South West Stockholm Psychiatry (TIPS) will be included.

Scores on Alcohol Use disorder identification Test (AUDIT) and Drug Use disorder Identification Test (DUDIT) will be used as a covariate in order to control for the patients' s drug and alcohol use habits.

The study is single blind randomized controlled trials of manualized Cognitive Behavior Group Therapy (CBGT) versus an active treatment condition of individual CBT for patients with first episode psychosis. A total of 16 patients are enrolled and randomly allocated to either CBGT or to individual CBT treatment. Then 18 structured CBGT or individual CBT sessions approximately once a week will be offered. Three experienced CBT trained therapists will perform the therapies. Two therapists will be allocated to each group composed by approximately 5 patients.

The group therapies are conducted according to the Acceptance and Commitment Therapy (ACT) for psychosis manual (an 18 Session Group Therapy Protocol by Pearson A. & Tingey R.). The individual therapies are conducted according to non-manualized ordinary clinical procedure. The ACT manual is originally constructed for patients with chronic schizophrenia and has therefore been adapted by the therapists to be appropriate for patients with first episode psychosis. The therapists have taken a course in ACT and they receive ACT-supervision during the trial.

Assessments in both studies will be carried out at baseline, after therapy completion and 6 months later by an independent rater blind to group allocation and not involved in the treatment of the patients. The raters blindness will be measured.

ELIGIBILITY:
Inclusion criteria: Diagnostic and Statistical Manual 5 (DSM-5):

* schizophrenia spectrum disorders:
* schizophrenia,
* schizophreniform psychosis,
* schizoaffective disorder)
* delusional disorder,
* brief psychotic disorder
* psychosis not otherwise classified.

Exclusion Criteria:

* Patients with drug abuse diagnosis
* organic brain injury,
* patients with grave somatic illness with secondary psychotic symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Symptoms of psychoses | Up to 11 months
  measured with PANSS (subscales: positive and negative symptoms).

SECONDARY OUTCOMES:
Quality of Life, | Up to 11 months
  Quality of life is measured by Brunnsviken Brief Quality of Life Inventory.
Symptoms of depression | Up to 11 months
  Symptoms of Depression; Becks Depression Inventory.
Self Esteem | Up to 11 months
  Self esteem is measured by Self Concept Questionaire
Values, | Up to 11 months
  Living in accordance with ones values is measured by Bull´s eye Values Survey.
Psychological inflexibility and Experiential Avoidance. | Up to 11 months
  Psychological inflexibility and experiential avoidance is measured with Acceptance and Action Questionaire II
Treatment safety | Up to 11 months
  Treatment safety is evaluated through assessment of adverse effects or events by registering suicide, suicide attempts, re-hospitalization and severe depressive symptom exacerbation).
Symptoms of anxiety | Up to 11 months
  Becks Anxiety Inventory,
Alcohol use | Upt to 11 months
  Alcohol Use Disorder Identification Test
Drug use | Up to 11 months
  Drug Use Disorder Identification Test.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Fatouros-Bergman, PhD, Principal Investigator — Karolinska Insitutet